CLINICAL TRIAL: NCT02800902
Title: Comparative Evaluation of Locally Delivered 1.2% Atorvastatin and 1.2% Rosuvastatin Gel in Treatment of Mandibular Degree ii Furcation Defects in Chronic Periodontitis Subjects: A Randomized Controlled Clinical Trial
Brief Title: Locally Delivered Atorvastatin & Rosuvastatin for Treatment of Furcation Defects in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and HOD, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2014-2015U8
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- group 1 (Placebo Comparator): Scaling and root planing (SRP) followed by placebo gel local drug delivery
  Interventions: Drug: placebo
- group 2 (Active Comparator): SRP followed by 1.2% rosuvastatin (RSV) gel
  Interventions: Drug: Rosuvastatin
- group 3 (Active Comparator): SRP followed by 1.2% Atorvastatin (ATV) gel
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: placebo — Oral prophylaxis followed by placement of placebo gel
  Other Names: inactive drug
  Arms: group 1
Drug: Rosuvastatin — Oral prophylaxis followed by placement of rosuvastatin gel
  Other Names: RSV
  Arms: group 2
Drug: Atorvastatin — Oral prophylaxis followed by placement of atorvastatin gel
  Other Names: ATV
  Arms: group 3

SUMMARY:
Statins are one of the lipid lowering drugs that help in reducing cholesterol levels in the body by specifically inhibiting 3-hydroxy-3-methylglutaryl coenzyme A reductase; which is a rate limiting enzyme for cholesterol synthesis. Rosuvastatin (RSV) and atorvastatin (ATV) have shown to have bone stimulatory and anti-inflammatory effects.. The present study aims to explore the efficacy of 1.2% RSV and 1.2% ATV gel as a local drug delivery and redelivery system as an adjunct to scaling and root planing (SRP) for the treatment of degree II furcation defects.

DETAILED DESCRIPTION:
Statins are one of the lipid lowering drugs that help in reducing cholesterol levels in the body by specifically inhibiting 3-hydroxy-3-methylglutaryl coenzyme A reductase; which is a rate limiting enzyme for cholesterol synthesis. Rosuvastatin (RSV) and atorvastatin (ATV) have shown to have bone stimulatory and anti-inflammatory effects.. The present study aims to explore the efficacy of 1.2% RSV and 1.2% ATV gel as a local drug delivery and redelivery system as an adjunct to scaling and root planing (SRP) for the treatment of degree II furcation defects.

Methods: Ninety patients with mandibular buccal class II furcation defects were randomly allocated into three treatment groups: SRP plus placebo gel (group 1), SRP plus 1.2% RSV gel (group 2) and 1.2% ATV gel (group3). Clinical and radiographic parameters were recorded at baseline then after 6 months. The gels were redelivered at the respective sites at this 6 month appointment. Then again all clinical and radiographic parameters were recorded after 3 months. (9 months from baseline)

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with mandibular class II furcation defects and asymptomatic endodontically vital mandibular molars with radiolucency in furcation area with PD ≥ 5mm and horizontal PD ≥ 3mm and with no history of antibiotic or any periodontal therapy in past 6 months were included in the study

Exclusion Criteria:

* Subjects with any known systemic disease, allergic to statins, on systemic statin therapy, alcoholics, tobacco users, pregnant or lactating women

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Bone defect fill | baseline, 6 & 9 months
  Assessed in percentage

SECONDARY OUTCOMES:
Change in modified sulcus bleeding index | baseline, 6 & 9 months
  scale 0-3
Change in Plaque index | baseline, 6 & 9 months
  scale 0-3
Change in pocket probing depth | baseline, 6 & 9 months
  measured in mm
Change in relative vertical clinical attachment level | baseline, 6 & 9 months
  measured in mm
Change in relative horizontal clinical attachment level | baseline, 6 & 9 months
  measured in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Garg S, Pradeep AR. 1.2% Rosuvastatin and 1.2% Atorvastatin Gel Local Drug Delivery and Redelivery in the Treatment of Class II Furcation Defects: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Mar;88(3):259-265. doi: 10.1902/jop.2016.160399. Epub 2016 Oct 7. PMID 27715376